CLINICAL TRIAL: NCT05917145
Title: Phase 0/I Clinical Trial of the ATM-Inhibitor WSD0628 in Combination With Radiation Therapy for Recurrent High-Grade Glioma
Brief Title: ATM-Inhibitor WSD0628 in Combination With Radiation Therapy for Treatment of Recurrent High-Grade Glioma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MC220712; R01FD007842 (FDA); 23-004794 (Other: Mayo Clinic Institutional Review Board); NCI-2023-06935 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2023-06-15; First posted 2023-06-23 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Intervention Model Description: Group A - Dose Escalation Phase Group B - Dose Expansion Group C - Tumor Penetrance Cohort
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group A (Dose Escalation) (Experimental): WSD0628 treatment should be started the day before radiation therapy starts (Day 1). Radiation therapy is given for 10 consecutive business days (Day 2-15, not including weekends and holidays), and WSD0628 will only be given on those 10 consecutive business days ≥30 minutes but ≤2 hours before radiation.
  Interventions: Drug: WSD0628
- Group B (Dose Expansion) (Experimental): WSD0628 treatment should be started the day before radiation therapy starts (Day 1). Radiation therapy is given for 10 consecutive business days (Day 2-15, not including weekends and holidays), and WSD0628 will only be given on those 10 consecutive business days ≥30 minutes but ≤2 hours before radiation.
  The Group B (Dose Expansion) portion of the study will be opened after the Group A (Dose Escalation) is complete.
  Interventions: Drug: WSD0628
- Group C (Tumor Penetrance Treatments) (Experimental): One treatment of WSD0628 will be given prior to radiation and surgical resection will be performed on the same day. The two doses given will be determined by Group A and Group B. Patients will be randomized in a 1:1 fashion.
  * Dose level 1: minimally radiosensitizing concentration of WSD0628 will be achieved.
  * Dose level 2: selected based on a prediction that a maximally radiosensitizing concentration of WSD0628 will be achieved.
  This portion of the study will open after Group A (Dose Escalation) is complete. This portion of the study will open to patients with recurrent high-grade glioma to further evaluate the efficacy, safety, tolerability, pharmacokinetics and biological activity of WSD0628 when combined with radiation therapy in specific patient subgroups
  Interventions: Drug: WSD0628

INTERVENTIONS:
Drug: WSD0628 — A non-toxic compound and inhibits the DNA damage response associated with radiation therapy. • WSD-0628 radio sensitizes Glioblastoma cells.

SUMMARY:
The purpose of this study is to test WSD0628 in combination with radiation therapy for recurrent brain tumors.

DETAILED DESCRIPTION:
High grade gliomas are the most common primary brain tumor in adults. Despite aggressive treatment including surgery, chemotherapy, and radiation, these tumors have a dismal prognosis. Following a radiation therapy, almost 80% of them recur locally. The focus of this project is the development of a radiation sensitizer (a small molecule ATM inhibitor, WSD0628) with the goal to enhance the efficacy of radiation therapy. The first step will be to establish a pre-clinical PK→PD→efficacy model to describe WSD0628 plasma and tumor concentrations associated with robust ATM inhibition and radiosensitizing effects. This model will be instrumental in interpreting the pharmacokinetic (PK) data and dosage selection in the proposed first-in-human, Phase 1, open-label, multicenter, single-arm, dose-escalation, and dose-expansion study in approximately 42 adult patients with recurrent high-grade glioma. The aims of the study are to assess the safety, tolerability, PKs and preliminary anti-tumor activity of WSD0628 in combination with radiation therapy. The dose-escalation portion of the study (Part A) will enroll approximately 24 patients and is comprised of Bayesian Optimal Interval (BOIN) design with target toxicity rate of 22%-33%. Once the recommended Phase 2 dose (RP2D) is established, Part B of the study will commence in which an additional 12 patients will be enrolled and treated at the RP2D for further evaluation of safety and efficacy (standard expansion cohort), and an additional 6 patients will have a tissue evaluation of tumor penetrance after a one-time dose of study drug prior to radiosurgery and surgical resection (Phase 0, tumor penetrance cohort). Tumor response will be assessed, using brain magnetic resonance imaging (MRI) with assessment based on the Response Assessment in Neuro-Oncology (RANO) criteria, and safety will include analysis of adverse events (AEs) and laboratory data. Additionally, PK, pharmacodynamic (PD), overall survival, progression-free survival, overall response rate, and patient-reported outcomes will be evaluated. The maximum duration of Part A will be 32 months and Part B,12 months. Funding Source - FDA OOPD

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Histological confirmation of one of the following:

  * Glioblastoma, IDH-wildtype
  * Grade 3 or 4 IDH1/2 mutant astrocytoma (2021 WHO classification)
  * Measurable disease as defined in Section 11.0
  * Disease progression after previous treatment for glioma with radiation and chemotherapy
* Minimum life expectancy of at least 3 months
* Group C only: Dose Expansion, Brain Tumor Penetration Group: plan for radiosurgery and surgical resection as part of routine clinical care
* ECOG Performance Status (PS) 0, 1 or 2 (Appendix I)
* The following laboratory values obtained ≤15 days prior to registration:

  * Hemoglobin ≥9.0 g/dL
  * Leukocytes ≥3.0 x 109/L
  * Absolute neutrophil count (ANC) ≥1500/mm3 or 1.5 x 109/L
  * Platelet count ≥100,000/mm3 or 100 x 109/L
  * Total bilirubin ≤1.5 x ULN and <3 mg/dL for patients with Gilbert's disease
  * Alanine aminotransferase (ALT) and aspartate transaminase (AST) ≤3 x ULN
  * PT/INR/aPTT ≤1.5 x ULN OR if patient is receiving anticoagulant therapy and INR or aPTT is within target range of therapy
* Calculated creatinine clearance ≥45 ml/min using the Cockcroft-Gault formula below:

  * Creatinine clearance for males = (140-age)(weight in kg)(72)(serum creatinine inmgdL⁄)
  * Creatinine clearance for females = (140-age)(weight in kg)(0.85)(72)(serum creatinine inmgdL⁄)
* Negative pregnancy test done ≤7 days prior to registration, for persons of childbearing potential only
* Willing to take light-protective measures during the study and for two weeks after their last dose of WSD0628
* Provide written informed consent
* Willing to return to enrolling institution for follow-up (during the Active Monitoring Phase of the study)
* Willingness to provide mandatory tissue specimens for correlative research

Exclusion Criteria:

* Any of the following because this study involves an investigational agent, the genotoxic, mutagenic, and teratogenic effects of which on the developing fetus and newborn are unknown:

  * Pregnant persons
  * Nursing persons
  * Persons of childbearing potential and persons able to father a child who are unwilling to employ adequate contraception
* Uncontrolled intercurrent illness including, but not limited to:

  * ongoing or active infection
  * symptomatic congestive heart failure
  * unstable angina pectoris
  * cardiac arrhythmia
  * or psychiatric illness/social situations that would limit compliance with study requirements
* Any of the following cardiac criteria:

  * Marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >480 milliseconds (ms) (CTCAE Grade 1) using Fredericia's QT correction formula.
  * History of additional risk factors for Torsades de Pointes (e.g., heart failure, hypokalemia, family history of Long QT. Syndrome).
  * Use of concomitant medications that prolong the QT/QTc interval
  * History of myocardial infarction ≤6 months prior to registration, or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias
* Known coagulopathy increasing the risk of bleeding or history of clinically significant hemorrhage, including significant intracranial tumor related hemorrhage
* Any of the following medications:

  * Enzyme-inducing anticonvulsants within two weeks of enrollment NOTE: Patients can be enrolled after a change to non-enzyme inducing anticonvulsants)
  * Patients taking more than 8 mg of dexamethasone per day (or equivalent steroid dose) at time of enrollment
* Any of the following prior therapies:

  * Radiation therapy <= 26 weeks prior to registration (including gamma tiles)
  * Chemotherapy, immunotherapy, or any investigational drug <= four weeks prior to registration,
  * or carmustine (BCNU) or lomustine (CCNU) <= six weeks prior to registration
* Past medical history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis which required steroid treatment, or any evidence of clinically active interstitial lung disease
* History of hypersensitivity to active or inactive excipients of WSD0628 or drugs with a similar chemical structure or class to WSD0628
* Refractory nausea and vomiting if not controlled by supportive therapy, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of WSD0628
* Uncontrolled hypertension
* History of severe brain-injury or stroke
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2024-01-17 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Determine the maximum tolerated dose of WSD0628 in combination with radiation therapy for patients with recurrent high-grade glioma. | 4 weeks after last day of RT (up to 60 days)
  Use Bayesian Optimal Interval (BOIN) design to inform dose escalation and de-escalation decisions and to ultimately determine the maximum tolerated dose level (MTD) of WSD0628 in patient population.
Determine the recommended phase 2 dose of WSD0628 in combination with radiation therapy for patients with recurrent high-grade glioma. | 4 weeks after last day of RT (up to 60 days)
  Evaluate biologic activity measures using rank-based desirability scores (RDS) generated for each of the dose levels to identify which of these scores best when looking jointly at toxicity and biologic activity. The rank-based desirability scores (RDS) for this BOIN12 design will be used to help identify the best dose

SECONDARY OUTCOMES:
Measure the incidence of acute adverse effects related to WSD0628 delivered concurrently with radiation | 4 weeks after last day of RT (up to 60 days)
  All AEs must be documented in the subject's medical record
Assess anti-tumor activity of WSD0628 delivered concurrently with radiation, including intracranial overall response rate (ORR) | 4 weeks after last day of RT (up to 60 days)
  Overall response rate defined as the proportion of patients who achieve a partial response (PR) or a complete response (CR) divided by the total number of patients who received therapy. Exact binomial 95% confidence intervals for the overall response rate will be calculated.
Assess anti-tumor activity of WSD0628 delivered concurrently with radiation, including progression-free survival (PFS) | Beginning of study therapy until the first occurrence of progression or death
  The primary measure of response will be by serial measures of the product of the two largest cross-sectional diameters (bidirectional product) using the RANO and iRANO criteria.
Assess anti-tumor activity of WSD0628 delivered concurrently with radiation, including volumetric change in tumor size | Beginning of study therapy until the first occurrence of progression or death
  measured by MRI/CT scan evaluations

CONTACTS AND LOCATIONS:
Overall Officials: William G. Breen, MD, Principal Investigator — Mayo Clinic; Jann N. Sarkaria, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials